CLINICAL TRIAL: NCT04091399
Title: Multi-centre, Open-label, First-in-man Study of Adult Patients Suffered From Alveolar Osteitis Treated Using Stomatological Tamponade Contipro
Brief Title: First-in-man Study of Adult Patients Suffered From Alveolar Osteitis Treated Using Stomatological Tamponade Contipro
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Contipro Pharma a.s. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PT-ST-1_12-14
Record Dates: First submitted 2019-09-08; First posted 2019-09-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Alveolar Osteitis
Keywords: first-man-study; alveolitis sicca dolorosa; alveolar osteitis; alveolalgia; sodium hyaluronate; octenidine hydrochlorid; clinical study
MeSH Terms: conditions — Dry Socket

STUDY DESIGN:
Intervention Model Description: 1. Collection personal data of patients suffered from alveolar osteotis
  2. Patient cohort selection according inclusion and exlusion criteria
  3. Extraction wound examination and characteriyation of a dry socket
  4. Treatment of alveolar osteoitis using a tested drug
  5. Extraction wound healing process and its evaluation
  6. Data analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient cohort (Experimental): Patients suffered from alveolar osteitis and treated using a Stomatological tamponade Contipro, composed of the Hyaluronic acid and Octenidine dihydrochloride. Firstly, the extraction wound had been irrigated with 2 ml of 3% solution of H2O2 to disinfect the site and then flushed by 2 ml of Aqua pro injectione to clear any remaining debris. After, the tested drug was applied into the extraction wound. This procedure was repeated on a daily basis for a maximum of 7 days or until the pain subsided below 20 mm and remained there for at least 2 days.
  Interventions: Drug: Stamatological tamponade Contipro

INTERVENTIONS:
Drug: Stamatological tamponade Contipro — The drug is composed from the Hyaluronic acid and Octenidine dihydrochloride. It is designed to perform comparatively in pain alleviation and to promote healing of the alveolar osteitis while avoiding the side effects.

SUMMARY:
Alveolar Osteitis (AO) is a complication following extraction of a tooth. AO manifests by localized pain in and around the extraction site where the postoperative blood clot has been disintegrated. The aim of this study was to determinate if there are any concerns of use of a pharmacological drug composed of an octenidine and lyophilized hyaluronic acid in a treatment of AO.

The tested drug is a sponge-like material composed solely of fully absorbable medicaments. It was designed to serve as non-toxic, slow-dissolving antiseptic which adheres to mucosa and so obturate the wound. The treatment was considered effective when the pain subsided to < 20mm VAS in < 8 days of treatment.

DETAILED DESCRIPTION:
Alveolar Osteitis (AO) is a complication following extraction of a tooth. AO manifests by localized pain in and around the extraction site where the postoperative blood clot has been disintegrated. The AO incidence is reportedly conditioned by multiple risk factors including trauma/difficult extraction, smoking, acute inflammation of periodontal tissues (e.g. dentitio difficilis) prior to extraction. The use of oral contraceptives results in about 10 times higher incidence of AO. Furthermore, secondary contributing risk factors include age, flap design, local anesthetic containing vasoconstrictor, and bone/root debris left in the extraction wound. The drug tested in this study was composed from the Hyaluronic acid (HA) and Octenidine dihydrochloride (ODC). It was designed to perform comparatively in pain alleviation and to promote healing while avoiding the side effects.

The aim of this clinical study was to determinate if there are any concerns of use a pharmacological drug composed of ODC and HA in treatment of AO. The drug was designed to fulfill the following criteria: to disinfect the wound (provided by ODC), attach to the mucosa (HA), obturate the wound (HA), be stable in the presence of saliva (HA), be fully absorbable (ODC, HA), enhance healing process (HA), be non-allergic and have analgesic effect (ODC, HA).

The sponge-like pharmacological drug is a lyophilized water solution of ODC, HA, stabilized with calcium chloride; as such it is fully dissoluble, has antiseptic properties and is malleable. The drug was manufactured by Contipro Pharma a.s. (Czech Republic). The study was designed as a multi-center, open-label, first-in-men study and was approved by the ethical committee of the University Hospital Hradec Králové.

Upon the study initiation, the study subjects' extraction wounds were examined and described by the medical professional and the subjects' perceived-pain self-evaluation base data was recorded. The perceived pain was recorded on 0-100 mm VAS. Afterwards, the treatment was introduced. Firstly, the wound had been irrigated with 2 ml of 3% solution of H2O2 to disinfect the site and then flushed by 2 ml of Aqua pro injectione to clear any remaining debris. After, the tested drug was applied into the extraction wound. This procedure was repeated on a daily basis for a maximum of 7 days or until the pain subsided below 20 mm and remained there for at least 2 days.

The treatment was considered effective when the pain subsided to < 20mm VAS in < 8 days of treatment. Descriptive statistics were provided for each of the criteria using the following values: 1) for continuous data: mean, standard deviation (SD), median, lower/upper quartile, minimum and maximum values, 2) for qualitative data: absolute count and percentages. Hypotheses are tested at standard cutoff α = 0.05.

A descriptive analysis approach (including frequency tables) was used to assess clinical management, clinical outcomes and healthcare resources used. When appropriate two-sided 95% confidence interval was obtained for population characteristics of a variable. All calculations and summaries were produced using R version 3.2.3 (R Core Team, Austria).

ELIGIBILITY:
Inclusion Criteria:

* Patient with diagnosed alveolar osteitis
* Minimal age limit 18 years
* Patient capable to fully understand and comply with the requirements of the study

Exclusion Criteria:

* Patient younger than 18 years
* Pregnant or lactant woman
* Patient diagnosed with cancer
* Patient with a history of radiotherapy in the head and neck area
* Patient undergone bisphosphonate treatment within the last two years
* Patient who had been given antibiotics less than two weeks prior the AO onset
* Patient with hypersensitivity or allergy to any substances contained in the tested drug
* Patient who smokes more than 10 cigarettes per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-09-11 (Actual); Primary Completion 2016-02-12 (Actual); Study Completion 2016-02-12 (Actual)

PRIMARY OUTCOMES:
The number of patients with treated related adverse effects objectively evaluated by examiners | 7 days/per patient
  The prevalence of potential treatment-relatived adverse effect evaluated by dentists in follow-up examinations

SECONDARY OUTCOMES:
Pain change assessed by the VAS scale according to subjective evaluation by patients | 7 days/per patient
  Pain change was assessed by the VAS scale. Pain relief associated with treatment was determinated as drop on the VAS scale below 20 mm

OTHER OUTCOMES:
Extraction wound healing assessed by objectively evaluation of examiners | 7 days/per patient
  Examinars evaluated the extraction wound healing as a change of inflammation of the impacted alveolae on scale 0 - 5 (0 - no inflammation, 5 - persistant inflammation).

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Suchánek, MUDr., Principal Investigator — University Hospital Hradec Králové
Locations (11):
- Czechia (11):
  - IchtysDent s.r.o, Brno
  - University Hospital Brno, Clinic of Oral, Maxillary and Facial Surgery, Brno
  - Prouzovi s.r.o., Dvůr Králové nad Labem
  - University Hospital Hradec Králové, Department of Dentistry, Hradec Králové
  - Dentine s.r.o., Jičín
  - FSmile s.r.o., Opočno
  - Dentpra, Pardubice
  - Mojmír Strnad, Pardubice
  - MEDIKAP, Pardubice
  - DV Dent s.r.o., Roudnice nad Labem
  - Enta Dent s.r.o, Ústí nad Labem

IPD SHARING:
Plan to Share IPD: No